CLINICAL TRIAL: NCT02457143
Title: Comparing Methods of Recall for Cancer Screening in Primary Care: a Pragmatic Randomized Clinical Trial
Brief Title: Comparing Methods of Recall for Cancer Screening in Primary Care: a Pragmatic Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15-145
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Early Detection of Cancer; Cancer; Socioeconomic Status
Keywords: recall; income-related disparities; cancer screening
MeSH Terms: conditions — Neoplasms | interventions — College Fraternities and Sororities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letter (Experimental): Patients will receive a reminder letter signed by their family physician which indicates which cancer screening tests they are overdue for and encourages them to book an appointment for screening.
  Interventions: Behavioral: Letter
- Phone call (Experimental): Patients will receive a phone call from a member of the practice staff. The call will inform them about which cancer screening tests they are overdue for and will encourage them to book an appointment for screening.
  Interventions: Behavioral: Phone call

INTERVENTIONS:
Behavioral: Letter
  Arms: Letter
Behavioral: Phone call
  Arms: Phone call

SUMMARY:
This randomized trial aims to understand how effective a reminder letter is compared to a reminder phone call in improving breast, cervical and colorectal cancer screening rates and reducing screening disparities.

ELIGIBILITY:
Inclusion Criteria:

* The trial will include patients who are rostered to the family practice as of March 31, 2015, are eligible and overdue for cervical, breast and/or colorectal cancer screening and are verified by their primary care physician as needing recall.

Exclusion Criteria:

* Patients will be excluded if their primary care physician noted they should not be recalled for screening or if the patient does not have both an address and a phone number on file.

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5270 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in each arm who go on to receive at least one screening test for which they are due | 6 months
The proportion of patients in each arm who are due for breast, cervical and colorectal cancer screening who go on to receive those respective screening tests (female patients may be represented in the outcome calculation of more than one cancer screening | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Lofters, MD PhD CCFP, Principal Investigator — Unity Health Toronto; Tara Kiran, MD MSc CCFP, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Academic Family Health Team, Toronto, Ontario, Canada